CLINICAL TRIAL: NCT06668350
Title: Racial/Ethnic Differences in Appeal and Preference for Flavored Little Cigars/Cigarillos: A Multi-Method Approach to Inform Tobacco Policy
Brief Title: Attitudes and Perceptions Attitudes and Smoking Perceptions in the Real Environment -II
Acronym: ASPIRE-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ACS CHERC; CHERC-24-1160021-01-CHERC (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cigarillo Flavor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Concept flavored cigarillo (Experimental): Participants will smoke a concept flavored cigarillo in the lab
  Interventions: Other: Smoking outcomes
- Characterizing flavored cigarillo (Experimental): Participants will smoke a characterizing flavored cigarillo
  Interventions: Other: Smoking outcomes
- Tobacco flavored cigarillo (Experimental): Participants will smoke a tobacco flavored cigarillo
  Interventions: Other: Smoking outcomes

INTERVENTIONS:
Other: Smoking outcomes — Participants will be assessed on several smoking outcomes including puffing behavior, subjective effects, and exhaled carbon monoxide

SUMMARY:
This multi-method project will recruit young adults who currently use cigarillos and examine the effects of different flavored cigarillo types (concept, characterizing, tobacco) on three measures of tobacco product appeal: subjective effects (e.g., taste, enjoyment, satisfaction, reward), actual smoking behavior (e.g., number of puffs), and tobacco product purchases via a simulated experimental tobacco marketplace.

ELIGIBILITY:
Inclusion Criteria:

* Ages18 to 34
* Smoke a little cigar or cigarillo (LCCs) "some days" or "everyday" (verified by brand name of the product);
* Ability to read English at an 8th grade level or higher; and
* No immediate plans to quit using tobacco
* > 1 prior experience, even 1 puff, with a flavored tobacco product
* U.S. Citizen or permanent resident of the United States.

Exclusion Criteria:

* Current use of nicotine replacement therapy (NRT) or stop smoking medication;
* Pregnant, planning to become pregnant, or currently breastfeeding;
* Past or current self-reported clinically significant heart disease or hypertension, or other smoking-related disease (by history) that preclude successful study completion;
* Inability to abstain from nicotine/tobacco products for at least 12 hours prior to lab sessions
* Report using the study cigarillo brand as their preferred brand (as this will likely unduly influence their perceptions)
* Unwillingness to use "untipped" (e.g., plastic or wood tip) little cigars/cigarillos.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Puff volume | From enrollment to the end of the study at 6 weeks
  Volume of inhaled cigarillo puffs
Subjective effects from smoking | From enrollment to the end of the study at 6 weeks
  Self-reported reward from cigarillo smoking from a questionnaire. This scale has 5 questions with response options ranging from 1 - not at all to 7 - extremely. The score is averaged across the number of items. Higher ratings indicate greater psychological reward.
Exhaled carbon monoxide | From enrollment to the end of the study at 6 weeks
  Changes in exhaled carbon monoxide (CO boot) following cigarillo smoking

CONTACTS AND LOCATIONS:
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided